CLINICAL TRIAL: NCT06743334
Title: Secondary Databased Post-marketing Surveillance Study of BNT162b2
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591056
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19 Vaccines; Safety; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; famtozinameran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- All primary series recipients using monovalent vaccine: All individuals who received first dose with monovalent vaccine as primary series (6 months or older).
  Interventions: Biological: Tozinameran (BNT162b2)
- First booster recipients with monovalent vaccine: All individuals who received first booster recipients with monovalent vaccine (5 years of age or older).
  Interventions: Biological: Tozinameran (BNT162b2)
- Second booster recipients with monovalent vaccine: All individuals who received second booster recipients with monovalent vaccine (5 years of age or older).
  Interventions: Biological: Tozinameran (BNT162b2)
- All booster recipients using bivalent vaccine: All individuals who received booster recipients using bivalent vaccine (12 years of age or older).
  Interventions: Biological: Tozinameran (BNT162b2) / Riltozinameran (BNT162b2 OMI BA.1); Biological: Tozinameran (BNT162b2) / Famtozinameran (BNT162b2 OMI BA.4-5)
- Single-dose primary series recipients with bivalent vaccine: All individuals who received single-dose primary series recipients with bivalent vaccine (12 years of age or older).
  Interventions: Biological: Tozinameran (BNT162b2) / Riltozinameran (BNT162b2 OMI BA.1); Biological: Tozinameran (BNT162b2) / Famtozinameran (BNT162b2 OMI BA.4-5)
- Primary series recipients with first dose of monovalent vaccine and second dose of bivalent vaccine: All individuals who received primary series recipients with first dose of monovalent vaccine and second dose of bivalent vaccine (12 years of age or older).
  Interventions: Biological: Tozinameran (BNT162b2) / Riltozinameran (BNT162b2 OMI BA.1); Biological: Tozinameran (BNT162b2) / Famtozinameran (BNT162b2 OMI BA.4-5)

INTERVENTIONS:
Biological: Tozinameran (BNT162b2) — 1. 12 years or older
     * Primary series: 2 doses, 30 μg each, administered 21 days apart
     * Booster shot (dose 3): 1 dose, 30 μg after ≥ 6 months from the second shot
  2. 5 to 11 years of age
     * Primary series: 2 doses, 10 μg each, administered 21 days apart
     * Booster shot (dose 3): 1 dose, 10 μg after ≥ 6 months from the second shot
  3. 6 months to 4 years of age
     * Primary series: 3 doses (2 doses of 3 μg each, administered 21 days apart, followed by 1 dose after ≥8 weeks)
  Groups: All primary series recipients using monovalent vaccine; First booster recipients with monovalent vaccine; Second booster recipients with monovalent vaccine
Biological: Tozinameran (BNT162b2) / Riltozinameran (BNT162b2 OMI BA.1) — 1. 12 years or older
  - Single booster dose, 15/15 μg, administered after ≥3 months after primary series
  Groups: All booster recipients using bivalent vaccine; Primary series recipients with first dose of monovalent vaccine and second dose of bivalent vaccine; Single-dose primary series recipients with bivalent vaccine
Biological: Tozinameran (BNT162b2) / Famtozinameran (BNT162b2 OMI BA.4-5) — 1. 12 years or older
  - Single booster dose, 15/15 μg administered after ≥3 months after primary series
  Groups: All booster recipients using bivalent vaccine; Primary series recipients with first dose of monovalent vaccine and second dose of bivalent vaccine; Single-dose primary series recipients with bivalent vaccine

SUMMARY:
This study is to assess the post-marketing safety of BNT162b2 products using nationwide population-based database in Republic of Korea.

DETAILED DESCRIPTION:
This study is a retrospective, non-interventional, observational study using Korean Disease Control and Prevention Agency-COVID-19-National Health Insurance Service (K-COV-N) database that includes COVID-19 vaccination/infection and claims data in Korean population. For the primary objective, cohort and self-controlled design will be used for measure of occurrence and measure of association, respectively. For the secondary objective, cohort design will be used for measure of occurrence.

Primary objective:

* To describe the frequency and estimate the incidence ratio of adverse events of special interest (AESIs) following exposure to Comirnaty Injection among individuals aged 6 months or older in the Republic of Korea
* To evaluate the relative risk of AESIs following exposure to Comirnaty Injection among individuals aged 6 months or older in the Republic of Korea, using a self-controlled case series (SCCS) design

Secondary objective:

- To describe the frequency and estimate the incidence ratio of severe COVID-19 outcomes (COVID-19 hospital admission, COVID-19 intensive care unit [ICU] admission, and COVID-19 death).

ELIGIBILITY:
1. Primary Objectives 1-1. Measure of Occurrence Inclusion Criteria For the measure of occurrence, analytical populations will include following individuals,

   * Who meet the predefined criteria for each study population.
   * With enrollment in the national insurance during the observation period, as well as during the clean window prior to the start of the observation period.

   Exclusion Criteria For the measure of occurrence, analytical populations will exclude following individuals,
   * With diagnosis of AESI during the AESI-specific clean window; or
   * With diagnosis of AESI between first dose and second/third dose of primary series when analyzing for the second/third dose.

   1-2. Measure of Association Inclusion Criteria For the measure of association, analytical populations will include following individuals,
   * Who meet the predefined criteria for each study population.
   * With enrollment in the national insurance during the observation period, as well as during the clean window prior to the start of the observation period; and
   * Who had incident AESI during the observation period. Exclusion Criteria For the measure of association, analytical populations will exclude following individuals,
   * Who do not have both risk and control window time. If an individual disenrolls, dies, or reaches the end of the study period during the risk window prior to accumulating any control window time, he/she will be excluded; or
   * With a diagnosis of AESI during the AESI-specific clean window.
2. Secondary Objective Inclusion Criteria For the secondary objective, the study populations will include following individuals,

   * Who meet the predefined criteria for each study population. Exclusion Criteria
   * None

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who were vaccinated with at least one dose of Pfizer COVID-19 vaccine according to locally approved label in Republic of Korea from 27 February 2021 through 31 December 2023.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events of Special Interest (AESI) - Measure of Occurrence | Up to 270 days after vaccination
  Measure of Occurrence (Cohort design) The frequency of AESIs will be analyzed.
Incidence of Adverse Events of Special Interest (AESI) - Measure of Occurrence | Up to 270 days after vaccination
  Measure of Occurrence (Cohort design) The incidence of AESIs will be analyzed.
Incidence of Adverse Events of Special Interest (AESI) - Measure of Association | Up to 270 days after vaccination
  Measure of Association (Self-Controlled Design) The incidence of AESIs will be analyzed.

SECONDARY OUTCOMES:
Frequency of Severe COVID-19 Outcomes | Up to 150 days after vaccination
  The frequency of severe COVID-19 outcomes including COVID-19 hospital admission, COVID-19 Intensive care unit (ICU) admission, and COVID-19 death will be estimated.
Incidence of Severe COVID-19 Outcomes | Up to 150 days after vaccination
  The incidence of severe COVID-19 outcomes including COVID-19 hospital admission, COVID-19 Intensive care unit (ICU) admission, and COVID-19 death will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.